CLINICAL TRIAL: NCT01391845
Title: Effect of Ulipristal Acetate Administration on Serum Progesterone Levels and Glycodelin-A Endometrial Pattern in Women Undergoing Controlled Ovulation Stimulation.
Brief Title: Ulipristal Acetate on Progesterone Levels and Glycodelin-A Endometrial Pattern
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Programa de Asistencia Reproductiva de Rosario (Other)
Responsible Party: Idelma Serpa, Programa de asistencia reproductiva de rosario (PROAR)
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: ist1979
Record Dates: First submitted 2011-06-28; First posted 2011-07-12 (Estimated); Last update posted 2011-07-20 (Estimated); Status verified 2011-05

CONDITIONS: Infertility
Keywords: progesterone; glycodelin-A; ulipristal acetate
MeSH Terms: conditions — Infertility | interventions — ulipristal acetate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- UPA, 300UI FSH (Experimental): patients on COS with 300UI FSHu/GnRH Antagonist protocol and ulipristal acetate use
  Interventions: Drug: ulipristal acetate
- No UPA, 300FSH (Placebo Comparator): patients on COS with 300UI FSHu/GnRH Antagonist protocol and without ulipristal acetate use
  Interventions: Drug: placebo
- UPA, FSH 225 (Experimental): patients on COS with 225UI FSHu/GnRH Antagonist protocol and ulipristal acetate use
  Interventions: Drug: ulipristal acetate
- no UPA, FSH225 (Placebo Comparator): patients on COS with 225UI FSHu/GnRH Antagonist protocol and without ulipristal acetate use
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: ulipristal acetate — 30mg of ulipristal acetate orally the day of hCG injection in a unique dose
  Other Names: UPA/FSH 300
  Arms: UPA, 300UI FSH
Drug: placebo — placebo orally in a unique dose the day of hCG injection
  Other Names: No UPA/FSH 300
  Arms: No UPA, 300FSH
Drug: ulipristal acetate — ulipristal acetate 30mg orally in a unique dose the day of hCG administration
  Other Names: UPA/FSH225
  Arms: UPA, FSH 225
Drug: placebo — placebo orally in a unique dose the day of hCG injection
  Other Names: no UPA/FSH225
  Arms: no UPA, FSH225

SUMMARY:
Controlled ovarian stimulation (COS) for FIV increases progesterone (P) and estradiol (E2) serum levels in supraphysiologic concentrations at the end of follicular phase. Elevated serum P levels leads to an accelerated endometrial maturation which interferes with the dialogue between embryo and endometrium. It has been reported that serum progesterone levels ≥ 1.5 ng/ml on the last day of COS are related to a significant decrease in the ongoing pregnancy rate following IVF cycles. Also, it has been reported a significant alteration in the endometrial gene expression profile related to P elevated levels.

Glycodelin-A is an immunomodulatory glycoprotein synthesized by luteal-phase endometrial epithelium and its expression seems to be related to the action of P. Because glycodelin-A has immunosuppressive activity, it may facilitate the process of implantation and the maintenance of pregnancy.

It is already know that ulipristal acetate (UPA) decrease serum P levels. The hypothesis of this study is that UPA is been able to modify P serum levels and glycodelin-A endometrial expression pattern on FSH/GnRH Antagonist cycles for FIV.

DETAILED DESCRIPTION:
Controlled ovarian stimulation (COS) for FIV increases progesterone (P) and estradiol (E2) serum levels in supraphysiologic concentrations at the end of follicular phase. Elevated serum P levels leads to an accelerated endometrial maturation which interferes with the dialogue between embryo and endometrium. It has been reported that serum progesterone levels ≥ 1.5 ng/ml on the last day of COS are related to a significant decrease in the ongoing pregnancy rate following IVF cycles. Also, it has been reported a significant alteration in the endometrial gene expression profile related to P elevated levels.

Glycodelin-A is an immunomodulatory glycoprotein synthesized by luteal-phase endometrial epithelium and its expression seems to be related to the action of P. Because glycodelin-A has immunosuppressive activity, it may facilitate the process of implantation and the maintenance of pregnancy.

Objective: to evaluate the endometrial effect of Progesterone through Glycodelin-A expression pattern on women exposed or not to ulipristal acetate in GnRH Antagonist cycles using two different doses of FSH for ovarian controlled stimulation.

Methods: prospective controlled randomized study. It will be enrolling 16 oocytes donors from Oocyte Donation Program of PROAR (a Reproductive Center of Rosario, Argentina). On day 3 of menstrual cycle FSH serum levels and antral follicular count (AFC) will be measure. If those results fulfill with inclusions criteria, patients will be randomize for FSH 225UI or 300UI GnRH-Antagonist/ urinary FSH protocol. P serum levels will be measure every 48 hours since at least 1 follicle ≥14 mm will be achieve until at least 1 follicle reach 19mm of diameter. The next day of hCG administration a new P circulating will be measure and then the patient will be randomize trough opaque envelopes for receive 30mg of ulipristal acetate or placebo. An endometrial biopsy with Cornier´s Pipelle will be performing 3 and 5 days after hCG injection (hCG+3 and hCG+5 days) to evaluate endometrial dating and Glycodelin-A expression pattern.

Statistical analysis: nominal variables will be analyzing using t-Student test and the effect of ulipristal with ANOVA.

ELIGIBILITY:
Inclusion Criteria:

* Age <35 years old
* FSH on day 3: <12 UI/ml
* Antral follicular count ≥ 6 on day 3 of the cycle
* BMI: <30 Kg/m2

Exclusion Criteria:

* Hypothyroidism
* Hyperprolactinemia
* Kidney or liver disease
* Smoking
* Alcoholism

Ages: 21 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2011-07; Primary Completion 2012-03 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Changes in Glycodelin-A endometrial expression pattern and Progesterone serum levels in women expose to ulipristal acetate on stimulated ovarian cycles for FIV | participants will be followed for the duration of one mesntrual cycle, from day 1 of the cycle until day 28-32
  to evaluate Glycodelin-A expression pattern by immunohistochemistry and Progesterone serum levels on women exposed or not to ulipristal acetate in FSH/GnRH Antagonist protocol.

SECONDARY OUTCOMES:
P levels during controlled ovarian stimulation since at least one follicle achieve ≥14mm of diameter | participants will be followed for the duration of one mesntrual cycle,from day 1 until day 28-32
Serum P levels on two different doses of FSH in a GnRH Antagonist protocol for ovarian stimulation | participants will be followed for the duration of one mesntrual cycle,from day 1 until day 28-32
Glycodelin-A endometrial expression pattern on two different doses of FSH in a GnRH Antagonist protocol for ovarian stimulation | participants will be followed for the duration of one mesntrual cycle, from day 1 until day 28-32

CONTACTS AND LOCATIONS:
Overall Officials: Idelma Serpa, MD, Principal Investigator — PROAR-IUNIR; Carlos Morente, MD, Study Chair — Programa de Asistencia Reproductiva de Rosario
Locations (1):
- PROAR (Programa de Asistencia Reproductiva de Rosario, Rosario, Santa Fe Province, Argentina